CLINICAL TRIAL: NCT05494060
Title: XELOX Combined With Anlotinib and Penpulimab vs XELOX as Adjuvant Therapy in ctDNA Positive Gastric and Esophagogastric Junction Adenocarcinoma, a Randomized, Controlled, Multicenter Clinical Trial
Brief Title: XELOX Combined With Anlotinib and Penpulimab vs XELOX as Adjuvant Therapy in ctDNA Positive Gastric and Esophagogastric Junction Adenocarcinoma
Acronym: EXPLORING
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-SR-342
Record Dates: First submitted 2022-08-08; First posted 2022-08-09 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Carcinoma; Gastrointestinal Diseases; Stomach Cancer; Gastroesophageal-junction Cancer; Digestive System Diseases; Gastric Cancer; Gastrointestinal Neoplasms
Keywords: Penpulimab; Anlotinib; Capecitabine; Oxaliplatin; ctDNA; adjuvant therapy
MeSH Terms: conditions — Carcinoma; Gastrointestinal Diseases; Stomach Neoplasms; Digestive System Diseases; Gastrointestinal Neoplasms | interventions — penpulimab; XELOX; Capecitabine; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Experimental: Penpulimab + Anlotinib + XELOX； Active Comparator: XELOX
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Penpulimab + Anlotinib + XELOX (Experimental): Penpulimab in combination with Anlotinib and XELOX (Capecitabine and Oxaliplatin)
  Interventions: Drug: Anlotinib hydrochloride capsule; Drug: Penpulimab Injection; Drug: XELOX
- XELOX (Active Comparator): XELOX (Capecitabine and Oxaliplatin)
  Interventions: Drug: XELOX

INTERVENTIONS:
Drug: Anlotinib hydrochloride capsule — Anlotinib hydrochloride capsule 12mg given orally in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21)；
  Arms: Penpulimab + Anlotinib + XELOX
Drug: Penpulimab Injection — Penpulimab Injection 100mg per bottle, 200mg IV Day 1, cycled every 21 days
  Other Names: AK-105
  Arms: Penpulimab + Anlotinib + XELOX
Drug: XELOX — Capecitabine:1000 mg/m2 bid d1-14 q3w, Oxaliplatin:130 mg/m2 d1 q3w
  Other Names: Capecitabine and Oxaliplatin

SUMMARY:
This is an open label, randomized, phase Ⅱ, multi-cohort study to treat subjects with ctDNA Positive Gastric and Esophagogastric Junction Adenocarcinoma. The patients will be randomized into two arms consist of Penpulimab + Anlotinib (3 weeks/cycle) + XELOX and XELOX at a ratio of 1:1. This study is conducted to assess safety and anti-tumor activity of the monoclonal antibody Penpulimab in combination with Anlotinib and standard chemotherapy as adjuvant treatment for ctDNA-positive Gastric, or Gastroesophageal Junction Carcinoma.

DETAILED DESCRIPTION:
This is an open label, randomized, phase Ⅱ, multi-cohort study to treat subjects with ctDNA Positive Gastric and Esophagogastric Junction Adenocarcinoma. The patients will be randomized into two arms consist of Penpulimab + Anlotinib (3 weeks/cycle) + XELOX and XELOX at a ratio of 1:1. This study is conducted to assess safety and anti-tumor activity of the monoclonal antibody Penpulimab in combination with Anlotinib and standard chemotherapy as adjuvant treatment for ctDNA-positive Gastric, or Gastroesophageal Junction Carcinoma. The study includes a screening (up to 28 days), treatment (disease recurrence, unacceptable toxicity, or subject withdrawal of consent with a maximum 12 month), safety follow-up (up to 30 days following last study drug treatment), and survival follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥18 and ≤75 years old, male or female.
* ECOG performance status score 0-1.
* Histologically or cytologically confirmed GC or GEJ carcinoma, had been treated with Radical resection (D2, R0 or R1) of gastric cancer.
* Pathological stage:III (8th AJCC TNM).
* Estimated lifetime is greater than 6 months.
* The main organs are functioning well, and the blood test results within 14 days before enrollment should meet the following requirements:

  1. Routine blood test:

     1. Hemoglobin (HB) ≥90 g/L.
     2. Neutrophil count (ANC) ≥1.5×109/L.
     3. Platelet count (PLT) ≥100×109/L.
  2. Biochemical test:

     1. Total bilirubin≤1.5×ULN (upper limit of normal).
     2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN; if there is liver metastasis, ALT and AST ≤ 5×ULN.
     3. Serum creatinine (Cr) ≤1.5 ULN or creatinine clearance ≥60mL/min.
* No obvious clinical symptoms of heart disease.
* Must have disease-free status documented by complete physical examination and imaging studies with no evidence of recurrent, residual, or metastatic disease on standard imaging (chest, abdomen, and pelvis captured by CT chest and CT or MRI of abdomen and pelvis) per investigator assessment within 28 days prior to enrollment.
* Females of childbearing potential must have a negative urine or serum pregnancy test within 7 days of randomization and must be willing to use a highly effective method of birth control (Appendix 9) for the duration of the study, and ≥ 120 days after the last dose of penpulimab and 180 days after the last dose of chemotherapy.
* Volunteer to participate in this study and sign an informed consent form.
* Considering that NGS analysis may take up to 10 working days, patients could receive 1 cycle of XELOX chemotherapy after ctDNA sampling.

Exclusion Criteria:

* Participation in other drug clinical trials within four weeks.
* Multiple factors affecting oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction.
* History of bleeding, any bleeding event with a severity grade of 3 or higher per CTCAE 5.0 within 4 weeks before screening.
* Patients with known central nervous system metastasis or history of central nervous system metastasis prior to screening. For patients with clinically suspected central nervous system metastases, CT or MRI must be performed within 28 days before enrollment to rule out central nervous system metastases.
* Patients with hypertension and uncontrolled by antihypertensive drugs alone (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg); Patients with a history of unstable angina pectoris; Patients newly diagnosed as angina pectoris within 3 months before screening or myocardial infarction events within 6 months before screening; Arrhythmias (including QTcF ≥ 450 ms in men, ≥ 470 ms in women requiring long-term use of antiarrhythmic drugs and New York Heart Association Class ≥ II cardiac insufficiency;There are many factors that affect oral drug absorption (such as inability to swallow, nausea and vomiting, upper gastrointestinal obstruction, abnormal physiological function, malabsorption syndrome, etc.), which may affect anlotinib hydrochloride absorbers.
* Long-term unhealed wound or unhealed fracture.
* Imaging findings show that the tumor has invaded around important blood vessels or the patient's tumor has a very high possibility of invading important blood vessels during treatment and causing fatal massive hemorrhage as judged by the investigator.
* Patients with abnormal coagulation function and bleeding tendency (the following criteria must be met within 14 days before randomization: INR is within normal range without anticoagulants or has no clinically significant abnormality); patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogues; patients with prothrombin time international normalized ratio (INR) ≤ 1.5 are allowed to take low-dose warfarin (1 mg orally, once daily) or low-dose aspirin (the daily dose does not exceed 100 mg) for preventive purposes.
* Arteriovenous thrombotic events occurred within 6 months before screening, such as cerebrovascular accident (including temporary ischemic attack), deep venous thrombosis (except venous thrombosis caused by previous chemotherapy that has been judged by the investigator to have recovered) and pulmonary embolism.
* Urine routine showed urine protein and 24 h urine protein was confirmed to be > 1.0g.
* Previous use of immune targeted therapy drugs.
* History of immunodeficiency, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation.
* Patients with infectious pneumonia, pneumonitis, interstitial pneumonia and other conditions requiring corticosteroids.
* History of severe chronic autoimmune diseases, such as systemic lupus erythematosus; history of inflammatory bowel disease such as ulcerative enteritis, Crohn's disease, irritable bowel syndrome and other chronic diarrheal diseases; history of sarcoidosis or tuberculosis; history of active hepatitis B, C and HIV infection; well-controlled non-serious immune diseases, such as dermatitis, arthritis, psoriasis, etc. Hepatitis B virus < 1000 copies/ml can be detected.
* Patients with hypersensitivity to human or murine monoclonal antibodies.
* Patients with a history of psychotropic substance abuse and unable to quit or with mental disorders.
* Pleural or peritoneal effusion with clinical symptoms requiring clinical intervention.
* Patients who do not follow the doctor's advice, do not take medicine as required, or have insufficient data that can affect the efficacy judgment or safety judgment.
* Patients with concomitant diseases that, in the judgment of the investigator, seriously jeopardize the patient's safety or affect the patient's completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | up to 2 years
  From date of receiving therapy until date of disease recurrence or death (by any cause in the absence of recurrence).

SECONDARY OUTCOMES:
Disease Free Survival (DFS) rate at 2 years | 2 years
  From date of receiving therapy until date of disease recurrence or death (by any cause in the absence of recurrence), assessed at 2 years.
Disease Free Survival (DFS) rate at 3 years | 3 years
  From date of receiving therapy until date of disease recurrence or death (by any cause in the absence of recurrence), assessed at 3 years.

OTHER OUTCOMES:
Overall survival (OS) | up to 4 years
  OS defined as the time from the first dose to death from any cause. Survival time was censored at the date of last contact for patients who were still alive or lost to follow-up.
Toxicity by CTCAE v5.0 criteria | up to 4 years
  oxicity and safety analysis will occur in patients who received at least one full or partial dose of study treatment. Adverse events will be graded per NCI CTCAE v.5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ext: Shu, PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen Y, Zhang J, Han G, Tang J, Guo F, Li W, Xie L, Xu H, Zhang X, Tian Y, Pan L, Shu Y, Ma L, Chen X. Efficacy and safety of XELOX combined with anlotinib and penpulimab vs XELOX as an adjuvant therapy for ctDNA-positive gastric and gastroesophageal junction adenocarcinoma: a protocol for a randomized, controlled, multicenter phase II clinical trial (EXPLORING study). Front Immunol. 2023 Oct 31;14:1232858. doi: 10.3389/fimmu.2023.1232858. eCollection 2023. PMID 38022553